CLINICAL TRIAL: NCT06558513
Title: Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Initial Efficacy of XNW5004 Tablets in Patients With Relapsed/Refractory Advanced Tumors
Brief Title: To Evaluate a Phase I/II Clinical Study of XNW5004 Tablets in Patients With Relapsed/Refractory Advanced Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW5004-I/II-01
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-08

CONDITIONS: Advanced Tumor; Lymphoma
Keywords: EZH2 inhibitor; XNW5004
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- XNW5004 (Experimental): Phase 1：treated with escalated doses of XNW5004 respectively； Phase 2：treated with RP2D of XNW5004 respectively
  Interventions: Drug: XNW5004 tablets

INTERVENTIONS:
Drug: XNW5004 tablets — XNW5004 an EZH2 inhibitor, BID, administered in continuous

SUMMARY:
Patients with advanced tumors diagnosed histologically or cytologically at the study center who were refractory to standard therapy or had relapsed received XNW5004 tablets

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old; Gender unlimited
* Pathologically confirmed, relapsed or refractory non Hodgkin's lymphoma (NHL). The definition of recurrence and refractory is as follows: Recurrence: After achieving remission, NHL meets the conditions for disease progression. For B-NHL patients, they should undergo a two line drug treatment regimen (with the first line containing CD20 monoclonal antibody), or a second line systemic treatment regimen that is not suitable/tolerated (such as toxic side effects, etc.); For T-NHL, first-line systemic chemotherapy should be administered, or if systemic chemotherapy is intolerant, and a regimen containing targeted CD30 drugs (including but not limited to Vibutuximab) or cetuximab should be administered. Refractory: Systemic medication treatment with at least two regimens and a total course of no less than 4 cycles of dose standard has not achieved partial remission.
* Only limited to stage IIa, pathologically diagnosed, relapsed or refractory follicular lymphoma, peripheral T-cell lymphoma, and diffuse large B-cell lymphoma, with recurrence and refractory defined according to inclusion criteria 2: Cohort 1: Follicular lymphoma (EZH2 mutant): Subjects whose genetic testing results showed the presence of EZH2 gene mutations; If the subject is unable to provide previous genetic testing results or there is no EZH2 gene mutation information in the previous genetic testing results, tumor tissue samples or bone marrow samples (only for subjects with bone marrow invasion) and blood samples must be provided. Only after confirming the presence of EZH2 gene mutations in the central laboratory can they be included in this queue; Cohort 2: Follicular lymphoma (EZH2 wild-type): subjects whose genetic testing results showed no EZH2 gene mutations; If the subject is unable to provide previous genetic testing results or there is no EZH2 gene mutation information in the previous genetic testing results, tumor tissue samples or bone marrow samples (only for subjects with bone marrow invasion) and blood samples must be provided. Only after confirmation by the central laboratory that there is no EZH2 gene mutation can they be included in this queue; Cohort 3: Peripheral T-cell lymphoma, according to the 2016 WHO classification of lymphoid tissue tumors; Cohort 4: Diffuse large B-cell lymphoma;
* At least one measurable lesion should be used as the evaluation basis
* During the dose escalation phase, subjects should provide tumor tissue samples or bone marrow samples (limited to subjects with bone marrow invasion) and oral swabs (control samples) as much as possible. If tumor tissue or bone marrow samples cannot be provided, they can be included in the study after evaluation by the researcher, provided that they meet other inclusion criteria;
* Has a life expectancy of ≥12 weeks;
* The ECOG score is 0-1;
* The functional reserve of important organs meets the following requirements: (1) Hematopoietic function: a) Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L (≥ 0.5 × 10^9/L for those with bone marrow infiltration) (G-CSF was not used within one week before the screening period blood routine examination, and long-acting white needle was not used within two weeks); b) Platelet count ≥ 75 × 10^9/L (≥ 50 × 10^9/L for those with bone marrow infiltration) (no platelet transfusion or TPO receptor agonist used within one week before the screening period blood routine examination); c) Hemoglobin ≥ 90 g/L (bone marrow infiltration requires ≥ 70 g/L) (no red blood cells were transfused or EPO was used within one week before the screening period blood routine examination); (2) Liver function: serum total bilirubin ≤ 1.5 x ULN (Gilbert's syndrome ≤ 3 ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN, ALT/AST ≤ 5 x ULN for patients with liver infiltration, and alkaline phosphatase ≤ 5 x ULN for patients with liver and/or bone infiltration; (3) Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance rate estimated based on Cockcroft Gault formula ≥ 60 mL/min (Cockcroft Gault formula, see Appendix 5 for details); (4) Left ventricular ejection fraction (LVEF) ≥ 50%; (5) International standardized ratio (INR) or plasma prothrombin time (PT) ≤ 1.5 x ULN, partial thromboplastin time (APTT) ≤ 1.5 x ULN.
* Non surgical sterilization or female patients of childbearing age, as well as male subjects whose partners are female of childbearing age, are required to use a medically approved contraceptive measure (such as an intrauterine device, contraceptive pill, or condom) within 6 months after the screening period and the end of the study treatment period; Non surgically sterilized female patients of childbearing age must have a negative serum HCG test within 7 days prior to enrollment in the study, and must be non lactating;
* Prior to conducting research specific procedures, provide a written informed consent form with a signature and date, and be able to comply with clinical visits and research related procedures.

Exclusion Criteria:

* Patients who have previously received treatment with drugs similar or related to the investigational drug pathway (such as EZH 1/2 or EZH2 inhibitors);
* Those who have received anti-tumor treatment in the early stage but have not recovered their toxicity (according to NCI-CTCAE 5.0, the toxicity has not recovered to ≤ 1 level). Other toxicities that the researchers believe do not affect the safety evaluation of the subjects, such as hair loss, are excluded;
* Have a history of other malignant tumors within the 5 years prior to enrollment and do not meet clinical cure criteria. The following cases are excluded: skin basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast intraductal carcinoma in situ and thyroid papillary carcinoma that can be treated locally and have been cured.
* Impaired heart function or clinically severe heart disease, including any of the following: (1) Acute myocardial infarction or unstable angina before first administration ≤ 6 months; (2) Congestive heart failure (New York Heart Association classification of heart function as III or IV); (3) Uncorrected severe arrhythmia and hypertension ≥ 150/100mmHg; (4) Extended QTc interval (defined as>450ms in males and>470ms in females) (Fredericia's formula); (5) Have a history of other major cardiovascular diseases (such as valve replacement surgery, coronary artery bypass grafting surgery, etc.).
* Severe systemic active infection;
* HIV positive and syphilis (Anti TB) positive individuals;
* HBsAg positive and HBV-DNA copy number higher than the normal upper limit of detection value; Or HBcAb positive and HBV-DNA copy number higher than the normal upper limit of detection value; HCV antibody is positive, and the copy number of HCV RNA is higher than the normal upper limit of the detection value;
* There is a history of COVID-19 vaccination within one month before the first administration of this test, and there is a history of other vaccines within three months before the first administration of this test;
* Subjects who are known to be allergic to the investigational drug or its active ingredients or excipients;
* Patients who have undergone major surgery within 4 weeks prior to the start of treatment or plan to undergo major surgery during this study period (excluding surgeries such as puncture or lymph node biopsy);
* The subject is unable to swallow, or has a history of active gastrointestinal inflammation, chronic diarrhea, known diverticulosis, or has undergone gastrectomy or gastric banding that affects drug absorption. But gastroesophageal reflux disease that has been treated with proton pump inhibitors is allowed (if there is no possibility of drug interaction);
* Subjects who took known CYP3A4 inhibitors/inducers within 14 days prior to the first administration (see Appendix 7 for details);
* History of having T-cell lymphoblastic lymphoma (T-LBL) or T-cell lymphoblastic leukemia (T-ALL);
* Any history of malignant myeloid tumors, including myelodysplastic syndrome (MDS), or abnormal detection indicators related to MDS or myeloproliferative tumors (MPN);
* Individuals with a history of abuse or drug use of psychotropic substances;
* It is known that the subjects have bleeding prone diseases such as von Willebrand's disease or hemophilia, or require long-term treatment with warfarin or other vitamin K antagonists (such as phenylpropanoid coumarin);
* Individuals who may not be able to complete this study due to other reasons or whom the researcher believes should not be included.
* Previously suffering from or accompanied by central nervous system disorders, including but not limited to: epilepsy, paralysis, stroke, severe brain injury, senile dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, mental illness, etc;
* The presence of central nervous system or testicular invasion;
* Stage IIa only: follicular lymphoma grade 3b, mixed histology, or follicular lymphoma histologically transformed into diffuse large B-cell lymphoma;
* Stage IIa only: Diffuse large B-cell lymphoma diagnosed by FISH testing with MYC, BCL-2, and/or BCL-6 rearrangement;
* Stage IIa only: mycosis fungoides, S é zary syndrome, and primary cutaneous enlarged T-cell lymphoma;
* Burkitt's lymphoma, a gray area lymphoma between diffuse large B-cell lymphoma and Burkitt's lymphoma, and a gray area lymphoma between diffuse large B-cell lymphoma and Hodgkin's lymphoma;
* Previously received organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLo HSCT);
* Auto-HSCT (autologous hematopoietic stem cell transplantation) was performed within 3 months prior to administration in this experiment;
* Immunosuppressants are being used, including but not limited to: cyclosporine, tacrolimus, etc. used within 2 weeks prior to administration in this trial; Within 7 days before administration, receive high-dose corticosteroids (prednisone with a daily dose greater than 10mg or equivalent doses of other corticosteroids);
* Received radiotherapy within 4 weeks prior to administration in this trial;
* Received anti-tumor treatments such as chemotherapy, targeted therapy, and anti-tumor traditional Chinese medicine within 4 weeks prior to administration in this trial;
* Received immunotherapy within 4 weeks prior to administration in this trial;
* Received CAR-T treatment within 12 weeks prior to administration in this trial;
* Those who have used any other clinical trial drugs within 4 weeks prior to the administration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (AEs)[Safety and Tolerability] | through study completion, an average of about 10 months
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of XNW5004 will be assessed.
Recommended phase 2 dose (RP2D) | 28 days since the date of first dose in phase 1
  Recommended phase 2 dose (RP2D) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of XNW5004.

SECONDARY OUTCOMES:
Time to peak (Tmax) | 28 days since the date of first dose
  Pharmacokinetics profile of a single dose and continuous medication of XNW5004 and its metabolite (plasma): Time to peak (Tmax) of plasma concentration
Maximum plasma concentration (Cmax) | 28 days since the date of first dose
  Pharmacokinetics profile of a single dose and continuous medication of XNW5004 and its metabolite (plasma): Maximum plasma concentration (Cmax)
Halflife (T1/2) | 28 days since the date of first dose
  Pharmacokinetics profile of a single dose and continuous medication of XNW5004 and its metabolite (plasma): Halflife (T1/2)
Objective response rate (ORR) | every 8 weeks through study completion, an average of about 10 months
  Assess the response rate of subjects to the treatment of XNW5004
Progression-free survival (PFS) | every 8 weeks through study completion, an average of about 10 months
  Assess the progression-free survival of the subjects after the treatment of XNW5004
Duration of Response (DoR) | every 8 weeks through study completion, an average of about 10 months
  Assess the duration of Response of the subjects after the treatment of XNW5004
Complete response rate (CRR) | every 8 weeks through study completion, an average of about 10 months
  Assess the Complete response rate of the subjects after the treatment of XNW5004
Partial response rate (PRR) | every 8 weeks through study completion, an average of about 10 months
  Assess the partial response rate of the subjects after the treatment of XNW5004
Disease control rate (DCR) | every 8 weeks through study completion, an average of about 10 months
  Assess the disease control rate of the subjects after the treatment of XNW5004
The correlation between potential biomarkers (including but not limited to EZH2 mutations, etc.) and therapeutic efficacy | every 8 weeks through study completion, an average of about 10 months
  Assess the correlation between potential biomarkers (including but not limited to EZH2 mutations, etc.) and therapeutic efficacy of the subjects after the treatment of XNW5004
H3K27me3 (H3 histone 27th lysine trimethylation)/H3 histone relative baseline change level | 28 days since the date of first dose
  Assess the H3K27me3 (H3 histone 27th lysine trimethylation)/H3 histone relative baseline change level of the subjects after the treatment of XNW5004

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Lugui, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences; QI Junyuan, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, China